CLINICAL TRIAL: NCT06098833
Title: Treatment of Neonatal Encephalopathy With Oral Sildenafil Suspension to Repair Brain Injury Secondary to Birth Asphyxia: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate Safety and Efficacy (Phase II Study)
Brief Title: Treatment of Neonatal Encephalopathy With Oral Sildenafil Suspension to Repair Brain Injury Secondary to Birth Asphyxia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pia Wintermark (Other)
Responsible Party: Sponsor-Investigator, Pia Wintermark, Associate Professor of Pediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SANE-03
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Neonatal Encephalopathy
Keywords: birth asphyxia; brain; hypoxic-ischemic encephalopathy; neonate; neuroprotection; neurorestoration; newborn; sildenafil
MeSH Terms: conditions — Asphyxia Neonatorum; Hypoxia-Ischemia, Brain | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sildenafil (Active Comparator): Sildenafil per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life (dose 1=2mg/kg/dose, dose 2=2.5mg/kg/dose, and doses 3-14=3mg/kg/dose)
  Interventions: Drug: Sildenafil
- Ora-Blend (Placebo Comparator): Ora-Blend per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life (dose 1=2mg/kg/dose, dose 2=2.5mg/kg/dose, and doses 3-14=3mg/kg/dose)
  Interventions: Drug: Ora-Blend

INTERVENTIONS:
Drug: Sildenafil — Sildenafil per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life (dose 1=2mg/kg/dose, dose 2=2.5mg/kg/dose, and doses 3-14=3mg/kg/dose)
  Arms: Sildenafil
Drug: Ora-Blend — Ora-Blend per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life (dose 1=2mg/kg/dose, dose 2=2.5mg/kg/dose, and doses 3-14=3mg/kg/dose)
  Arms: Ora-Blend

SUMMARY:
Around the time of birth, some babies experience a condition called asphyxia, which means that their brain and other organs do not receive enough blood and/or oxygen to work properly. This life-threatening condition accounts for nearly 1 out of 4 deaths of all babies around the world, and often leads to severe brain damage, cerebral palsy, epilepsy, and trouble with learning and functioning in everyday life. At this time, no treatment is available to repair the brain damage caused by asphyxia. Excitingly, a drug called sildenafil (Viagra®) is already given safely to babies who suffer from increased blood pressure in their lungs' vessels. Recent studies using a laboratory model of asphyxia at birth suggest that sildenafil may also repair the brain damage caused by asphyxia. Similarly, recent small studies have shown that it is both feasible and safe to give sildenafil to human babies, who suffered from asphyxia at birth. These studies also highlight the first promising signs that sildenafil may improve how the brains of these babies work, which is consistent with the abovementioned laboratory studies.

On the basis of these previous researches, the investigators predict that sildenafil can repair the damage to a baby's brain. The investigators will test whether sildenafil can be safely given to a large group of human babies who suffer from asphyxia at birth, and will confirm whether sildenafil improves or not how their brains and hearts/lungs work.

This project will enable to determine whether sildenafil is a promising treatment for repairing brain damage in babies who suffer from asphyxia at birth. This project may also provide new solutions for these babies to improve their future life.

DETAILED DESCRIPTION:
The investigators will enroll neonates with HIE treated with TH from NICUs in a multicentre, randomized, double-blind, placebo-controlled phase 2 clinical trial to evaluate the safety and efficacy of sildenafil to repair brain injury. Neonates with moderate-severe HIE on admission and with brain injury on a day-2 brain MRI (during TH) will be randomized to sildenafil or placebo (allocation 2:1) for 7 consecutive days.

Aim 1: Evaluate the efficacy of sildenafil to improve brain injury (primary outcome). The investigators will determine whether sildenafil reduces brain injury on a day-30 MRI compared to the baseline day-2 MRI.

Aim 2: Determine the safety of sildenafil (secondary outcome). The investigators will assess the safety of sildenafil by recording the incidence of adverse events.

Aim 3: Evaluate the efficacy of sildenafil to improve cardiopulmonary hemodynamics (secondary outcome). The investigators will determine whether sildenafil improves pulmonary pressure and right/left ventricular function on day 4 of life (after TH completion) compared to baseline day-2 measurements

ELIGIBILITY:
Inclusion Criteria:

* Male and female neonates meeting the criteria for induced hypothermia:
* Gestational age ≥36weeks and birth weight ≥1800g;
* Evidence of fetal distress, i.e., history of an acute perinatal event, cord pH ≤7.0 or base deficit

  * 16 mEq/L;
* Evidence of neonatal distress, such as an Apgar score ≤5 at 10 minutes, postnatal blood gas pH obtained within the first hour of life ≤ 7.0 or base deficit ≤ - 16 mEq/L, or a continued need for ventilation initiated at birth and continued for at least 10 minutes;
* Evidence of moderate to severe neonatal encephalopathy by an abnormal neurological exam and/or an amplitude-integrated electroencephalogram (aEEG). They will receive whole-body cooling to an esophageal temperature of 33.5°C, initiated within the first 6 hours of life, continued for 72 hours, and then they will be slowly rewarmed using standard protocol.
* Evidence of brain injury on a brain magnetic resonance imaging (MRI) performed on day 2 of life.

Exclusion Criteria:

* Neonates with complex congenital heart disease
* Neonates with cerebral malformations
* Neonates with genetic syndrome
* Neonates with intraventricular and/or intraparenchymal hemorrhage on MRI performed on day 2 of life
* Moribund infants not expected to survive

Ages: 0 Minutes to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Extent of brain injury | Day 30 of life, compared to day 2 of life
  Primary outcome to explore efficacy (brain injury)

SECONDARY OUTCOMES:
Serious adverse events | Day 1 to 10 of life
  Close monitoring for adverse events such as death, hypotension, persistent pulmonary hypertension, altered renal or hepatic function, etc to assess the safety of sildenafil

OTHER OUTCOMES:
Ejection fraction (EF) in % (reflecting left ventricular function) and tricuspid annular plane systolic excursion (TAPSE) in cm (reflecting right ventricular function) | Day 2 to 4 of life
  Secondary outcome to explore efficacy (cardiopulmonary hemodynamics)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Wintermark, MD, Principal Investigator — Research Institute of the McGill University Health Centre (The Institute)
Locations (2):
- Canada (2):
  - Montreal Children's Hospital, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Related Info — http://www.neobrainlab.org